CLINICAL TRIAL: NCT01817296
Title: Klinefelter Syndrome: Are we Missing the Optimal Time for Fertility Preservation?
Brief Title: Klinefelter Fertility Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4093
Record Dates: First submitted 2013-03-13; First posted 2013-03-25 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Klinefelter Syndrome
Keywords: Klinefelter; Fertility
MeSH Terms: conditions — Klinefelter Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental)
  Interventions: Procedure: Testicular Biopsy

INTERVENTIONS:
Procedure: Testicular Biopsy — Micro-dissection testicular sperm extraction for sperm retrieval

SUMMARY:
Klinefelter syndrome occurs in 1 in 600 males and is a common cause of infertility in men. It appears scar tissue forms in these boys' testicles, leading to progressive destruction over their lifetimes. Advanced reproductive technology can be used to surgically retrieve sperm from these individuals, but these methods have a 50% failure rate in adult Klinefelter patients. Younger men have higher success rates, suggesting that adolescence and young adulthood may be the best time to extract sperm, but these techniques have not been studied in Klinefelter patients younger than 26 years of age. Additionally, there is currently no way to predict which Klinefelter patients will have success with these methods and which of them will not. This trial will explore sperm extraction in Klinefelter syndrome in an age range (12-25 years) that has never been studied, with the ultimate hope of improving the potential for fertility in these patients. The specific goals of this study are to determine the ideal age for sperm retrieval in Klinefelter patients and to establish factors that can be used to predict which of these patients will have a higher likelihood of success with advanced reproductive technology. The hypothesis is that younger Klinefelter patients will have higher sperm retrieval rates.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed 47,XXY (Klinefelter syndrome)
* 12-25 years of age

Exclusion Criteria:

* testosterone therapy within past 6 months
* history of surgery, injury, or infection in the testicle
* solitary testicle

Ages: 12 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Sperm retrieval rates based on age | Assessed at the end of the 6 month study period
  Results of testicular biopsies will be reviewed for each patient during the 6 month study period

SECONDARY OUTCOMES:
Correlation between sperm retrieval rates and physical and biochemical markers | Assessed at the end of the 6 month study period
  Results of testicular biopsies will be correlated to physical and biochemical markers for each patient after all of the data have been collected, during the 6 month study period.
Correlation between sperm retrieval rates and neurocognitive survey data | Assessed at the end of the 6 month study period
  Results of testicular biopsies will be correlated to neurocognitive survey data for each patient after all of the data have been collected, during the 6 month study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Nahata L, Yu RN, Paltiel HJ, Chow JS, Logvinenko T, Rosoklija I, Cohen LE. Sperm Retrieval in Adolescents and Young Adults with Klinefelter Syndrome: A Prospective, Pilot Study. J Pediatr. 2016 Mar;170:260-5.e1-2. doi: 10.1016/j.jpeds.2015.12.028. Epub 2015 Dec 31. PMID 26746120